CLINICAL TRIAL: NCT00269854
Title: A Placebo-Controlled, Dose-Ranging Study Followed by a Placebo-Controlled, Repeated-Dose Extension of Anti-TNF Chimeric Monoclonal Antibody (cA2) in the Treatment of Patients With Active Crohn's Disease
Brief Title: An Efficacy and Safety Study of Anti-TNF Monoclonal Antibody in Patients With Crohn's Disease
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Centocor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR006256
Record Dates: First submitted 2005-12-22; First posted 2005-12-26 (Estimated); Last update posted 2014-11-04 (Estimated); Status verified 2014-11

CONDITIONS: Crohn Disease
Keywords: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Infliximab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Infliximab 5 mg/kg (Experimental)
  Interventions: Drug: Infliximab 5 mg/kg
- Infliximab 10 mg/kg (Experimental)
  Interventions: Drug: Infliximab 10 mg/kg
- Infliximab 20 mg/kg (Experimental)
  Interventions: Drug: Infliximab 20 mg/kg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Infliximab 5 mg/kg — Infliximab (anti-TNF chimeric monoclonal antibody [cA2]) 10 milligram per kilogram (mg/kg) will be administered as infusion at Week 0, 2 and 6.
  Other Names: anti-TNF chimeric monoclonal antibody (cA2)
  Arms: Infliximab 5 mg/kg
Drug: Infliximab 10 mg/kg — Infliximab (anti-TNF chimeric monoclonal antibody [cA2]) 5 mg/kg will be administered as infusion at Week 0, 2 and 6.
  Other Names: anti-TNF chimeric monoclonal antibody (cA2)
  Arms: Infliximab 10 mg/kg
Drug: Infliximab 20 mg/kg — Infliximab (anti-TNF chimeric monoclonal antibody [cA2]) 20 mg/kg will be administered as infusion at Week 0, 2 and 6.
  Other Names: anti-TNF chimeric monoclonal antibody (cA2)
  Arms: Infliximab 20 mg/kg
Drug: Placebo — Matching placebo will be adminstered at Week 0, 2 and 6.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of anti-TNF chimeric monoclonal antibody (cA2) compared to placebo in patients with active Crohn's disease.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, double-blind, dose-ranging study followed by a placebo-controlled, double-blind, repeated-dose extension to evaluate the effectiveness and safety of anti-TNF chimeric monoclonal antibody (cA2) compared to placebo in the treatment of patients with active Crohn's disease. The primary efficacy outcome of the study is a comparison of the proportion of patients achieving a clinical response at the 4-week evaluation. Clinical response is defined as a reduction from baseline in the Crohn's Disease Activity Index (CDAI) score of at least 70 points. Additional measurements of effectiveness include the clinical response over time, the time to loss of response, clinical remission over time, and changes in the Crohn's Disease Activity Index (CDAI), Inflammatory Bowel Disease Questionnaire (IBDQ), Crohn's Disease Endoscopic Index of Severity (CDEIS) scores and C-reactive protein values.

Anti-TNF Chimeric Monoclonal Antibody (cA2) or placebo

ELIGIBILITY:
Inclusion Criteria:

* Patients with Crohn's disease of at least 6 months duration, with colitis, ileitis, or ileocolitis confirmed by radiography or endoscopy
* Having a Crohn's Disease Activity Index (CDAI) of >=220 and <=400
* Treated with at least 1 of the following: current use of oral corticosteroid therapy of <=40 mg/day (prednisone equivalent), current use of (or lack of response to) >=2 g/day of sulfasalazine (or equivalent) or >=800 mg of mesalamine, current use of (or lack of response to) azathioprine or 6-mercaptopurine, failure to respond to methotrexate or cyclosporine, (with a stop date at least 3 months prior to screening)
* If using oral corticosteroids, sulfasalazine or mesalamine, a start date at least 8 weeks prior to screening, with a stable dose of sulfasalazine or mesalamine for at least 4 weeks prior to screening and a stable dose of oral corticosteroids for at least 2 weeks prior to screening
* If not currently using oral corticosteroids, a stop date of any previous corticosteroid regimen of at least 4 weeks prior to screening and if not using sulfasalazine, mesalamine, azathioprine or 6-mercaptopurine, a stop date of any previous treatment with these agents of at least 8 weeks prior to screening

Exclusion Criteria:

* Patients with Crohn's disease limited to the stomach or proximal small intestine
* Having symptomatic stenosis or ileal strictures that might have require surgical intervention or that might render patients unresponsive to cA2 treatment
* Who have received treatment with parenteral corticosteroid or adrenocorticotrophic hormone within 4 weeks prior to screening, or currently requiring oral or parenteral corticosteroid therapy for another disease such as asthma
* Having a serious infection, such as hepatitis, pneumonia or pyelonephritis in the 3 months prior to screening, a history of opportunistic infection such as herpes zoster within 2 months prior to screening, or evidence of active cytomegalovirus, active pneumocystis carinii, or drug resistant atypical mycobacterium
* Having active signs or symptoms of severe, progressive or uncontrolled renal, hepatic, hematologic, endocrine, pulmonary, cardiac, neurologic or cerebral disease, or any current known malignancy or any history of malignancy which would put the patient at an unacceptable risk for participation in the study or that would be expected to limit life expectancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 1995-06; Primary Completion 1996-10 (Actual); Study Completion 1996-10 (Actual)

PRIMARY OUTCOMES:
Comparison of the proportion of patients achieving a clinical response at Week 4 | Week 4
  Clinical response is defined as a reduction from baseline in the Crohn's Disease Activity Index (CDAI) score of at least 70 points.

SECONDARY OUTCOMES:
Clinical response over time; Time to loss of response; Clinical remission over time; Changes in CDAI, Inflammatory Bowel Disease Questionnaire (IBDQ) and Crohn's Disease Endoscopic Index of Severity (CDEIS) scores and C-reactive protein values | up to Week 48

CONTACTS AND LOCATIONS:
Overall Officials: Centocor, Inc. Clinical Trial, Study Director — Centocor, Inc.

REFERENCES:
- [Result] Targan SR, Hanauer SB, van Deventer SJ, Mayer L, Present DH, Braakman T, DeWoody KL, Schaible TF, Rutgeerts PJ. A short-term study of chimeric monoclonal antibody cA2 to tumor necrosis factor alpha for Crohn's disease. Crohn's Disease cA2 Study Group. N Engl J Med. 1997 Oct 9;337(15):1029-35. doi: 10.1056/NEJM199710093371502. PMID 9321530